CLINICAL TRIAL: NCT06713317
Title: A Phase I Study to Evaluate the Safety and Drug Allergy of HLB3-002 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huonslab Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HLB3-002_P1
Record Dates: First submitted 2024-11-26; First posted 2024-12-03 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Healthy
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part I 'HLB3-002' (Experimental): Recombinant Hyaluronidase
  Interventions: Drug: HLB3-002
- Part I '0.9%NaCl' (Experimental): 0.9% Normal Saline
  Interventions: Drug: 0.9% NaCl
- Part II 'HLB3-002' (Experimental): Recombinant Hyaluronidase
  Interventions: Drug: HLB3-002
- Part II '0.9%NaCl' (Experimental): 0.9% Normal Saline
  Interventions: Drug: 0.9% NaCl

INTERVENTIONS:
Drug: HLB3-002 — Recombinant Hyaluronidase
  Arms: Part I 'HLB3-002'; Part II 'HLB3-002'
Drug: 0.9% NaCl — 0.9% Normal saline
  Arms: Part I '0.9%NaCl'; Part II '0.9%NaCl'

SUMMARY:
Part I) multi-center, randomized, double-blind, placebo controlled

Part II) multi-center, randomized, double-blind, placebo controlled

ELIGIBILITY:
Inclusion Criteria:

[Part I]

1. Healthy volunteers aged 19 years or older at the time of screening (Visit 1).
2. Subjects with intact skin at the site of administration, without tattoos, acne, dermatitis, pigmentation, or lesions that could interfere with the administration of the investigational drug and allergy testing.

[Part II]

1. Subjects who tested negative on the drug allergy assessment after Part 1 intradermal administration.
2. For women of childbearing potential, a negative pregnancy test (serum-hCG) at baseline visit (V5).

Exclusion Criteria:

[Part I]

1. Subjects with the following comorbidities or conditions:

   * Acute fever exceeding 37.5°C within 1 week prior to the baseline (Visit 2).
   * Symptoms of an acute illness within 2 weeks prior to the baseline (Visit 2).
   * Immune disorders that may affect the immune system (e.g., flu, cancer, HIV).
   * Chronic urticaria, dermographism.
   * Clinically significant diseases affecting the liver, kidneys, gastrointestinal system, cardiovascular system, respiratory system, endocrine system, immune system, psychiatric/neuropsychiatric system, hematologic system, or oncology.
   * Clinically significant blood pressure abnormalities.

     * Hypertension: Systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg.
     * Hypotension: Systolic blood pressure ≤90 mmHg and/or diastolic blood pressure ≤60 mmHg.
2. Subjects who have smoked more than 10 cigarettes per day within 4 weeks prior to the screening (Visit 1).
3. Subjects who have participated in another clinical trial and received investigational drugs or medical devices within 6 months prior to the baseline (Visit 2).
4. Other subjects deemed inappropriate for participation in this clinical trial by the investigator.

[Part II]

1) Subjects with the following comorbidities or conditions:

* Acute fever exceeding 37.5°C within 1 week prior to the baseline (Visit 5).
* Symptoms of an acute illness within 2 weeks prior to the baseline (Visit 5).
* Clinically significant diseases affecting the liver, kidneys, gastrointestinal system, cardiovascular system, respiratory system, endocrine system, immune system, psychiatric/neuropsychiatric system, hematologic system, or oncology.
* Clinically significant blood pressure abnormalities.

  * Hypertension: Systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg.
  * Hypotension: Systolic blood pressure ≤90 mmHg and/or diastolic blood pressure ≤60 mmHg.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Incidence rate of drug allergy following intradermal injection of the IP | 2 days
  Subject developing allergic reaction are considered to have drug allergy.

SECONDARY OUTCOMES:
Incidence rate of drug allergy following subcutaneous injection of the IP | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Donghoon Lee, MD, Ph.D, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No